CLINICAL TRIAL: NCT01671150
Title: Inflammation-Induced Depressed Mood: The Role of Social Neurocognitive Mechanisms
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Naomi Eisenberger, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Endotoxin 2; R01MH091352 (NIH)
Record Dates: First submitted 2012-07-11; First posted 2012-08-23 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Depression
Keywords: inflammation; depression; social cognition; neural activity
MeSH Terms: conditions — Depression; Inflammation | interventions — Endotoxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo control (Placebo Comparator): half of the participants will receive a placebo control
  Interventions: Drug: endotoxin
- Endotoxin (Inflammatory challenge) (Active Comparator)
  Interventions: Drug: endotoxin

INTERVENTIONS:
Drug: endotoxin — Low-dose endotoxin (0.8 ng/kg of body weight): EC.O:113 administered once

SUMMARY:
Depressive disorders occur at a high rate in patients with inflammatory disorders, with a point prevalence of 15-29%, which is two to three times greater than that observed in the general population. Substantial evidence has shown that inflammation and increases in proinflammatory cytokine activity play a critical role in the onset and perpetuation of depression and depressive symptoms (e.g. insomnia, fatigue) in those who are co-morbid for inflammatory disorders. Consistent with this, experimental work has shown that an inflammatory challenge can increase depressed mood in an otherwise healthy sample. Based on these findings, there has been a growing interest in whether inflammatory processes can contribute to depression in a causal manner and how these effects might occur.

Given the observation that inflammatory processes trigger social withdrawal, coupled with evidence that feelings of 'social disconnection' play a critical role in the onset and perpetuation of (non-inflammatory forms of) depression, it is surprising that the social psychological consequences of inflammation and their contribution to depression have not been more fully explored. Here, we suggest that inflammation may increase feelings of social disconnection and that these social psychological changes may be an important contributor to inflammation-associated depression. Indeed, preliminary data demonstrated that an experimentally-induced inflammatory challenge (endotoxin) led to increases in self-reported feelings of social disconnection (e.g., "I feel disconnected from others") in addition to increases in depressed mood. Aside from these findings, however, there are no studies that have explored the effect of inflammatory processes on social experience in humans. The over-arching objective of this proposal is to explore the experiential and neural correlates of inflammatory-induced changes in social experience (e.g., feelings of social disconnection), which may provide a critical missing link in understanding the relationship between inflammation and depression.

Participants (n=100) will be randomly assigned to receive either endotoxin or placebo and will then be monitored for the next six hours. Blood draws to assess cytokine levels as well as self-reported feelings of social disconnection and depressed mood will be collected hourly. In addition, at the time of peak cytokine response, participants will complete a neuroimaging session to examine the effect of inflammatory challenge on neural sensitivity to social rejection and social acceptance. It is hypothesized that endotoxin will increase feelings of social disconnection over time, and that the underlying neural sensitivities that give rise to these feelings (e.g., increased neural sensitivity to social rejection; decreased neural sensitivity to social acceptance) will contribute to inflammatory-induced depressed mood.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be required to be in good general health (as evaluated during the phone and in-person screening sessions described below), and to be between 18-50 years of age. All participants will be required to be fluent in English and to be right-handed.

Exclusion Criteria:

* Following a structured telephone interview, prospective participants with the following conditions will not advance to the in-person screening session: claustrophobia or presence of metal in their body (relevant for the neuroimaging component of the study), pregnant or planning to become pregnant in the next 6 months, presence of chronic mental or physical illness, history of allergies, autoimmune, liver, or other severe chronic diseases, current and regular use of prescription medications, nightshift work or time zone shifts (> 3hrs) within the previous 6 weeks, or previous history of fainting during blood draws.

Furthermore, the absence of significant health problems or medication use history will be confirmed by an in-person screening session. Any participant who has any of the following conditions will be ineligible for the study: Medical conditions. (1) presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders; (2) presence of co-morbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders; (3) presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk; (4) presence of chronic infection, which may elevate proinflammatory cytokines; (5) presence of an acute infectious illness in the two weeks prior to an experimental session. Psychiatric Disorders. (6) current and/or lifetime history of a major Depressive Disorder or other DSM-IV psychiatric disorder (e.g. substance dependence) due to the known effects of major depression and/or substance dependence on inflammation. (Absence of a psychiatric diagnosis will be based on a structured psychiatric interview (Structured Clinical Interview for DSM-IV Diagnosis: SCID; First et al., 1996).) Medication and substance use. (7) current and/or past regular use of hormone-containing medications including steroids; (8) current and/or past regular use of non-steroid anti-inflammatory drugs; (9) current and/or past regular use of immune modifying drugs that target specific immune responses such as TNF antagonists; (10) current and/or past regular use of analgesics such as opioids; (11) current and/or past regular use of psychotropic medications, including selective serotinergic reuptake inhibitors, antidepressants, anxiolytics, hypnotics, sedatives and barbiturates. Health factors. (12) current smokers or excessive caffeine users (>600 mg/day) because of known effects on proinflammatory cytokine levels; (13) body mass index (BMI) greater than 35, (14) shows evidence of drug use from a positive urine test, (15) has a positive pregnancy test, if female, or (16) shows any abnormalities on screening laboratory tests.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in depressed mood from baseline | at baseline and then at 1,2,3,4,5,and 6 hours after drug administration

SECONDARY OUTCOMES:
Neural activity to negative and positive social feedback | 2 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Eisenberger, PhD, Principal Investigator — University of California, Los Angeles; Michael Irwin, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Clinical & Translational Research Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Kruse JL, Boyle CC, Olmstead R, Breen EC, Tye SJ, Eisenberger NI, Irwin MR. Interleukin-8 and depressive responses to an inflammatory challenge: secondary analysis of a randomized controlled trial. Sci Rep. 2022 Jul 24;12(1):12627. doi: 10.1038/s41598-022-16364-3. PMID 35871638
- [Derived] Moieni M, Muscatell KA, Jevtic I, Breen EC, Irwin MR, Eisenberger NI. Sex Differences in the Effect of Inflammation on Subjective Social Status: A Randomized Controlled Trial of Endotoxin in Healthy Young Adults. Front Psychol. 2019 Oct 1;10:2167. doi: 10.3389/fpsyg.2019.02167. eCollection 2019. PMID 31632316
- [Derived] Moieni M, Tan KM, Inagaki TK, Muscatell KA, Dutcher JM, Jevtic I, Breen EC, Irwin MR, Eisenberger NI. Sex Differences in the Relationship Between Inflammation and Reward Sensitivity: A Randomized Controlled Trial of Endotoxin. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Jul;4(7):619-626. doi: 10.1016/j.bpsc.2019.03.010. Epub 2019 Apr 3. PMID 31103547
- [Derived] Moieni M, Irwin MR, Jevtic I, Breen EC, Cho HJ, Arevalo JM, Ma J, Cole SW, Eisenberger NI. Trait sensitivity to social disconnection enhances pro-inflammatory responses to a randomized controlled trial of endotoxin. Psychoneuroendocrinology. 2015 Dec;62:336-42. doi: 10.1016/j.psyneuen.2015.08.020. Epub 2015 Aug 28. PMID 26360770
- [Derived] Moieni M, Irwin MR, Jevtic I, Breen EC, Eisenberger NI. Inflammation impairs social cognitive processing: A randomized controlled trial of endotoxin. Brain Behav Immun. 2015 Aug;48:132-8. doi: 10.1016/j.bbi.2015.03.002. Epub 2015 Mar 10. PMID 25770082